CLINICAL TRIAL: NCT01780636
Title: Ultrasound and EMG Guided Botox Injection for the Treatment of Non-Relaxing Puborectalis Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: POOR RECRUITMENT
Sponsor: Karen Noblett (Other)
Collaborators: American Urogynecologic Society (Other); Allergan (Industry)
Responsible Party: Sponsor-Investigator, Karen Noblett, Professor of Obstetrics & Gynecology, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLERGAN-72570 HS# 2012-8750
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Non-relaxing Puborectalis Syndrome
Keywords: Non relaxing puborectalis syndrome; Botulinum toxin A; Botox; Constipation
MeSH Terms: conditions — Constipation | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulinum toxin (Botox) injection (Experimental): All patients will be given the active Botox injection and thus this study will remain open-label and non-randomized as this is a pilot study to determine initial efficacy.
  Interventions: Drug: botulinum toxin

INTERVENTIONS:
Drug: botulinum toxin
  Other Names: Botox (Allergan, Irvine, CA)

SUMMARY:
Our study aims to determine the efficacy of ultrasound and EMG guided Botox injections into the puborectalis muscle in women with non-relaxing puborectalis syndrome. With use of this technique, we believe we will find that Botox injections decrease symptom severity and improve quality of life (QOL) in patients with NRPS. All enrolled patients will receive ultrasound and EMG guided Botox injections at three points along the puborectalis muscle. Post-injection data will be obtained with a defecation diary and questionnaire data at the 2-week, 3-month, and 6-month intervals.

DETAILED DESCRIPTION:
Non-relaxing puborectalis syndrome (NRPS) is an obstructive defecatory disorder that presents with chronic constipation, anismus, or a sensation of incomplete rectal emptying. The specific etiology of this syndrome is unknown. The true incidence of NRPS is unknown, but it is estimated that 4% of patients with defecatory disorders have NRPS. Previous therapies for non-relaxing PRS have included biofeedback, pelvic floor physical therapy, dietary changes, laxatives, enemas, and surgical division of the puborectalis muscle. Unfortunately, responses to these treatments have been variable at best. Direct injection of botulinum toxin (Botox) into the puborectalis muscle is an alternative approach for treating NRPS and has recently been reported in a limited number of studies. Botox blocks cholinergic nerve endings in the autonomic nervous system and has been used to weaken the puborectalis muscle in constipated patients.

Our study aims to determine the efficacy of ultrasound and EMG guided Botox injections into the puborectalis muscle in women with NRPS. With use of this technique, we believe we will find that Botox injections decrease symptom severity and improve quality of life (QOL) in patients with NRPS.

We plan to compare patient reported symptoms, symptom severity, and QOL prior to Botox injections with symptoms and QOL at 2-week, 3-month, and 6-month intervals after Botox injection into the puborectalis muscle in patients with NRPS.

All enrolled patients will receive ultrasound and EMG guided Botox injections at three points along the puborectalis muscle. Post-injection data will be obtained with a defecation diary and questionnaire data at the 2-week, 3-month, and 6-month intervals. Additional injections will be offered to patients who fail the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Diagnosis of non-relaxing puborectalis syndrome

Exclusion Criteria:

* Allergy or sensitivity to botulinum toxin
* Pregnancy or plan to become pregnant in the subsequent 6 months after injection
* Undiagnosed ano-rectal mass, lesion, or infection
* Stage II or greater rectocele

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Times ML, Reickert CA. Functional anorectal disorders. Clin Colon Rectal Surg. 2005 May;18(2):109-15. doi: 10.1055/s-2005-870892. PMID 20011350
- [Background] WASSERMAN IF. PUBORECTALIS SYNDROME (RECTAL STENOSIS DUE TO ANORECTAL SPASM). Dis Colon Rectum. 1964 Mar-Apr;7:87-98. doi: 10.1007/BF02616902. No abstract available. PMID 14128302
- [Background] Kuijpers HC, Bleijenberg G. The spastic pelvic floor syndrome. A cause of constipation. Dis Colon Rectum. 1985 Sep;28(9):669-72. doi: 10.1007/BF02553449. PMID 4053909
- [Background] Karlbom U, Hallden M, Eeg-Olofsson KE, Pahlman L, Graf W. Results of biofeedback in constipated patients: a prospective study. Dis Colon Rectum. 1997 Oct;40(10):1149-55. doi: 10.1007/BF02055160. PMID 9336109
- [Background] Meunier P, Marechal JM, de Beaujeu MJ. Rectoanal pressures and rectal sensitivity studies in chronic childhood constipation. Gastroenterology. 1979 Aug;77(2):330-6. PMID 447047
- [Background] MacDonald A, Shearer M, Paterson PJ, Finlay IG. Relationship between outlet obstruction constipation and obstructed urinary flow. Br J Surg. 1991 Jun;78(6):693-5. doi: 10.1002/bjs.1800780620. PMID 2070237
- [Background] Mellgren A, Bremmer S, Johansson C, Dolk A, Uden R, Ahlback SO, Holmstrom B. Defecography. Results of investigations in 2,816 patients. Dis Colon Rectum. 1994 Nov;37(11):1133-41. doi: 10.1007/BF02049817. PMID 7956583
- [Background] Wexner SD, Jorge JM. Colorectal physiological tests: use or abuse of technology? Eur J Surg. 1994 Mar;160(3):167-74. PMID 8003569
- [Background] Halligan S, Malouf A, Bartram CI, Marshall M, Hollings N, Kamm MA. Predictive value of impaired evacuation at proctography in diagnosing anismus. AJR Am J Roentgenol. 2001 Sep;177(3):633-6. doi: 10.2214/ajr.177.3.1770633. PMID 11517060
- [Background] Salzano A, Cavallo G, De Rosa A, De Luca LE, Serpe A, Losco M. [Diagnosis with defecography of puborectal muscle syndrome]. Radiol Med. 1997 Apr;93(4):396-400. Italian. PMID 9244917
- [Background] Ganeshan A, Anderson EM, Upponi S, Planner AC, Slater A, Moore N, D'Costa H, Bungay H. Imaging of obstructed defecation. Clin Radiol. 2008 Jan;63(1):18-26. doi: 10.1016/j.crad.2007.05.015. Epub 2007 Sep 14. PMID 18068787
- [Background] Maria G, Brisinda G, Bentivoglio AR, Cassetta E, Albanese A. Botulinum toxin in the treatment of outlet obstruction constipation caused by puborectalis syndrome. Dis Colon Rectum. 2000 Mar;43(3):376-80. doi: 10.1007/BF02258305. PMID 10733120
- [Background] Maria G, Cadeddu F, Brandara F, Marniga G, Brisinda G. Experience with type A botulinum toxin for treatment of outlet-type constipation. Am J Gastroenterol. 2006 Nov;101(11):2570-5. doi: 10.1111/j.1572-0241.2006.00791.x. Epub 2006 Oct 4. PMID 17029615
- [Background] Ron Y, Avni Y, Lukovetski A, Wardi J, Geva D, Birkenfeld S, Halpern Z. Botulinum toxin type-A in therapy of patients with anismus. Dis Colon Rectum. 2001 Dec;44(12):1821-6. doi: 10.1007/BF02234461. PMID 11742168
- [Background] Shafik A, El-Sibai O. Botulin toxin in the treatment of nonrelaxing puborectalis syndrome. Dig Surg. 1998;15(4):347-51. doi: 10.1159/000018630. PMID 9845612
- See also: American Urogynecologic Society — http://www.augs.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Females over 18 were recruited from the URO/GYN and colorectal clinic. They have been diagnosed with non relaxing puborectalis syndrome.
Groups:
- Botulinum Toxin (Botox) Injection: All patients will be given the active Botox injection and thus this study will remain open-label and non-randomized as this is a pilot study to determine initial efficacy.
  botulinum toxin
Period: Overall Study
Arm/Group | Botulinum Toxin (Botox) Injection
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin (Botox) Injection
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: YEARS] | 55 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms Based on Scores Using the PAC-SYM and Wexner Constipation Questionnaires.
Description: To assess whether Botox injections into the puborectalis muscle will improve patient's symptoms based on scores using the PAC-SYM and Wexner Constipation validated questionnaires from baseline to 6 months post-Botox injection to determine severity of symptoms. The PAC-SYM questionnaire unabbreviated title is Patient Assessment of Constipation-Symptoms and the total score is summed ranging from 0 to 44. The Wexner Constipation questionnaire total score is summed ranging from 0 to 30. Both questionnaires have higher values representing a worse outcome.
Time Frame: Baseline to 6 months post-injection
Population: All females between the ages of 40-75 and data was insufficient to analyze as target enrollment was not met and terminated due to poor recruitment. The data for this outcome measure was not collected.
Arm/Group | Botulinum Toxin (Botox) Injection
Number analyzed (Participants) | 0

2. Primary Outcome: PAC-SYM and Wexner Scores
Description: Scores on a scale The baseline scores were compared to scores at 6 months to evaluate the degree of improvement
Time Frame: Baseline to 6 months
Population: All 7 received Botox and data was insufficient to analyze as target enrollment was not met and terminated due to poor recruitment. The data for this outcome measure was not collected.
Arm/Group | Botulinum Toxin (Botox) Injection
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Pressures on Anal Manometry
Description: To assess the change in pressures on anal manometry before and after Botox injections into the puborectalis muscle from baseline to 6 months post-Botox injection. Anal manometry is a test done in clinic to assess bowel function. Average resting pressure is recorded using the advanced diagnostic equipment. Above 40 mmHg is normal for resting pressure. Also, average squeeze pressure will be recorded. Greater than 100 mmHg is normal for average squeeze pressure.
Time Frame: Baseline to 6 months post-injection
Population: All female between ages 40-75. Data was insufficient to analyze as target enrollment was not met and terminated due to poor recruitment. The data for this outcome measure was not collected.
Arm/Group | Botulinum Toxin (Botox) Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition of adverse events did not differ from clinical trials.gov adverse events were monitored/assessed by the primary investigator
Arm/Group | Botulinum Toxin (Botox) Injection
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No